CLINICAL TRIAL: NCT03340129
Title: A Phase II, Open Label, Randomised, Controlled Trial of Ipilimumab and Nivolumab With Concurrent Intracranial Stereotactic Radiotherapy Versus Ipilimumab and Nivolumab Alone in Patients With Melanoma Brain Metastases.
Brief Title: Anti-PD 1 Brain Collaboration + Radiotherapy Extension (ABC-X Study)
Acronym: ABC-X
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma Institute Australia (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIA2019/CT/258 and CA209-8TJ; CA209-8TJ (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2017-08-28; First posted 2017-11-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Melanoma Stage Iv
Keywords: Immunotherapy; Radiotherapy; Brain metastases; Stereotactic radiotherapy; Stereotactic radiosurgery; Cognitive function; Neurological-specific cause of death
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Ipilimumab; Nivolumab; Radiosurgery; Salvage Therapy

STUDY DESIGN:
Intervention Model Description: Open label, randomised trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nivolumab + ipilimumab (Active Comparator): Nivolumab 1mg/kg and ipilimumab 3mg/kg Q3W x 4 doses, then nivolumab 480 mg every 4 weeks.
  Any form of salvage therapy (surgery or radiotherapy) may be administered to either cohort for the treatment of intracranial disease progression.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Other: Salvage therapy
- Nivolumab + ipilimumab,concurrent SRS (Active Comparator): Nivolumab 1mg/kg and ipilimumab 3mg/kg Q3W x 4 doses, then nivolumab 480 mg every 4 weeks.
  Stereotactic radiotherapy 16 to 22 Gy in 1 fraction or 24 to 30 Gy, hypofractionated for larger lesions. Stereotactic radiotherapy to commence within 7 days of of the baseline / planning MRI brain. Hypofractionated stereotactic radiotherapy should be completed within 14 day of the first fraction.
  Any form of salvage therapy (surgery or radiotherapy) may be administered to either cohort for the treatment of intracranial disease progression.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Radiation: Stereotactic Radiotherapy; Other: Salvage therapy

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 3mg per kg every 3 weeks for 4 doses
  Other Names: Yervoy
Drug: Nivolumab — Nivolumab 1mg/kg every 3 weeks for 4 doses, then 480mg every 4 weeks.
  Other Names: Opdivo
Radiation: Stereotactic Radiotherapy — The first dose of immunotherapy Must be given prior to the start of radiotherapy. One fraction at between 16 to 22 Gy or 24 to 30 Gy hypofractionated for larger lesions.
  Arms: Nivolumab + ipilimumab,concurrent SRS
Other: Salvage therapy — Any form of salvage therapy (surgery or radiotherapy) for intracranial disease progression, further disease control at any site, symptom control or treatment of cerebral haemorrhage or cerebral radionecrosis.

SUMMARY:
This is a phase II, open label, randomised trial of ipilimumab and nivolumab with concurrent intracranial stereotactic radiotherapy versus ipilimumab and nivolumab alone in patients with asymptomatic, untreated melanoma brain metastases.

DETAILED DESCRIPTION:
1. BACKGROUND The ABC study (NCT02374242) is a phase II clinical trial recruiting 3 cohorts of patients with melanoma brain metastases. 76 patients received immunotherapy with either nivolumab alone or nivolumab combined with ipilimumab. Nivolumab together with ipilimumab was shown to be more effective than nivolumab alone in melanoma brain metastases. The combination will therefore be used in this trial.

   Findings from pre-clinical and clinical research provides evidence supporting the ability of radiotherapy to induce anti-tumour immune responses and augment the efficacy of anti-PD1 checkpoint blockade in melanoma and provide mechanistic rationale for combined therapy.
2. STUDY DESIGN This current protocol builds on the ABC study and will assess clinical, functional, toxicities and quality of life outcomes with the combined modalities of immunotherapy with radiotherapy to the brain in melanoma patients.

   The main aim of this study will be to assess the effect of immunotherapy +/- concurrent stereotactic radiotherapy (SRS) on the intracranial death rate at 12 months from the commencement of treatment. Secondary aims include the RECIST response in the brain, extracranially and overall, progression free survival, overall survival, neurocognitive function, adverse event rates and quality of life.

   The study will recruit 218 patients with asymptomatic, untreated melanoma brain metastases. All patients will be treated with combination ipilimumab and nivolumab at the doses and duration approved by worldwide regulatory authorities for advanced melanoma. All patients will undergo the the SRS treatment planning MRI of the brain PRIOR to randomisation to ensure that the timing of the baseline intracranial measurements are made within a similar timeframe and so that the delineation of tumour volume is accurately recorded in the same way for both cohorts. Patents will be randomised to receive concurrent intracranial SRS (within 7 days of the baseline / planning MRI scan) or immunotherapy alone. At intracranial disease progression, any form of salvage local therapy (radiotherapy or surgery) may be administered to either cohort.

   Randomisation is 1:1, using a permuted, random block design with stratification by participating centre, LDH (normal / elevated), BRAF (mutant / wild type), 1-2 brain metastases versus > 2 brain metastases.
3. PRIMARY OUTCOME The neurological specific death rate at 12 months - defined as a proximate cause of death which is a sign, symptom, or diagnosis related to metastatic brain disease.
4. OBJECTIVE RESPONSES A modified version of RECIST will be used to assess response to treatment. The modification allows for up to 5 brain metastastes to be selected as target lesions and a further 5 extracranial lesions. The immune related response criteria (irRC) will also be applied and concordance evaluated with RECIST. The irRC measures the volume of tumour lesions by calculating bi-dimensional measurements of target lesions.
5. NEUROCOGNITIVE ASSESSMENT, FUNCTION AND QUALITY OF LIFE Neurocognitive impairment is a concern in the setting of radiotherapy delivered for brain metastases. The addition of immunotherapy for enhanced local disease control and survival may augment the risks. Quality of life (QoL) assessment is therefore an important objective in clinical trials studying the effects of new interventions, where side effects and tolerability are as important as clinical benefit.

   Neurocognitive function will be assessed at baseline and every 6 to 12 weeks using the Montreal Cognitive Assessment (MoCA) and a neurological assessment of the patient. A member of the study team will be nominated to conduct the MoCA to allow for consistency of delivery of the examination. The MoCA measures six cognitive domains: visuospatial/executive function; naming; memory; language; abstraction; and attention. To decrease the learning effect from multiple administrations of the MoCA over a short period of time, alternate versions have been made available.

   The Functional Assessment of Cancer Therapy (FACT) questionnaires are commonly used to assess cancer-related QoL issues. The FACT-Brain (FACT-Br) module provides an additional set of disease-specific questions pertaining to brain neoplasms and is completed by the patient.

   Neurological assessments wil be made using the structured NANO scale at each physical examination - each neurological domain is subdivided into 3 or 4 levels of function with scores based on discrete quantifiable measures. Thus, levels of function for each domain range from 0 to 2 or 0 to 3. A score of 0 indicates normal function, while the highest score indicates the most severe level of deficit for that domain. Levels of function are distinguished by significant and measurable differences in order to avoid misinterpretation of subtle or nonspecific changes.

   The EORTC QLQ-C30, an internationally validated cancer-specific QOL-instrument, assesses various facets of functioning, symptoms common in cancer patients and global QOL. The Brain Cancer Module (EORTC QLQ-BN20 is a 20-item supplement for the QLQ-C30 to assess neurological related quality of life and neurological symptoms and is being utilised in the main ABC study. Among the symptoms captured by neurocognitive tests are communication deficits and memory problems. In these cases, a patient-rated QoL tool may not capture the true effects of the disease or the intervention to treat it. Both C30 and BN20 modules have been validated for assessing health-related quality of life and symptoms in patients with brain cancer.

   General health status will also be measured using the EQ-5D. The EQ-5D is a standardized instrument for use as a measure of self-reported health status. The EQ-5D comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety) and a visual analogue rating scale (VAS). The utility data generated from the EQ-5D is commonly used in cost effectiveness analyses.
6. TOXICITY AND TOLERABILITY Adverse events will be reported using the CTCAE version 5.0 in addition to causality, duration, treatment required and the need for treatment delays or discontinuation. Radionecrosis is an event of clinical interest and will be captured separately.
7. CORRELATIVE BLOOD AND TISSUE BIOMARKER STUDIES Some patients may not benefit from radiation therapy and immunotherapy combinations. Therefore, biomarkers predictive of response. or the lack of it are needed. Extensive correlative analyses of tumoural and peripheral blood immunologic changes will be essential to a better understanding of the mechanistic interactions between these 2 treatment modalities. The differential composition of the gut microbiome has been shown to affect antitumor immunity and immunotherapy efficacy and will also be correlated with response and toxicity.

   To address this, blood, tissue, stool and urine samples will be obtained. Blood will be collected at baseline, at 1 week of treatment and then 6 to 12 weekly to examine serum chemokines, cytokines, inflammatory markers, lymphocyte and T cell subsets and myeloid derived suppressor cells and to assess correlation with disease response or progression. All Cohorts will be included in this study.

   In patients with sufficient archival melanoma tissue from metastatic sites, a baseline tumour PD-L1 level, immune markers and genetics of response and resistance will also be measured. If available, tumour tissue following progression of accessible extracranial disease and / or craniotomy will also be tested for immune and genetic markers.

   Stool samples will be obtained at baseline, at weeks 6 and 12 and at the end of immunotherapy to investigate the gut microbiome composition, diversity and abundance and correlation with the response to immunotherapy and immune-related gastrointestinal toxicity. A baseline evaluation of participants' dietary habits will also be included in these analyses.

   A reduction in intestinal barrier function is currently believed to play an important role in pathogenesis of many diseases, response to immunotherapy and immune related toxicity. Urinary excretion of two orally-administered non-metabolizable sugars, lactulose and mannitol, is a valuable marker for evaluating intestinal permeability. Patients will collect a urine specimen at baseline to assess this biomarker.
8. CONTINUED SYSTEMIC TREATMENT IN CASES OF PROGRESSIVE DISEASE

   The application of traditional RECIST criteria (Response Evaluation Criteria In Solid Tumors) in patients treated with immunotherapy may lead to premature discontinuation of treatment in a patient who will eventually respond to treatment or have prolonged disease stabilization. Disease progression may occur in extracranial lesions whilst patients may continue to have disease stabilisation or response of their intracranial melanoma disease, and vice versa. The patterns of response to treatment with these immunotherapy agents differ from those with molecularly targeted agents or cytotoxic chemotherapy in several important respects:
   * Patients may have a transient worsening of disease, manifested either by progression of known lesions or the appearance of new lesions, before disease stabilizes or tumour regresses. Therefore caution should be taken in abandoning therapy early. In general these delayed responses are not observed in patients with rapidly progressive, symptomatic disease.
   * Responses can take appreciably longer to become apparent compared with cytotoxic therapy. Continued disease regression is frequently observed well after completion of the initial induction period.
   * Some patients who do not meet traditional criteria for objective response can have prolonged periods of stable disease that are clinically significant.

   An evaluation of data from ipilimumab phase II clinical trials in advanced melanoma found patients characterized as PD at week 12 (by WHO criteria), either by an increase in tumour burden and/or the appearance of new lesions, subsequently experienced an objective response or SD (relative to baseline) without the addition of non-ipilimumab anticancer therapy. Examination of biopsies taken from patients receiving ipilimumab demonstrated that in some small unmeasurable lesions noted at baseline, an increase in size may be interpreted as PD, when instead, this may be due to inflammation due to T cell infiltration.
9. CONTINUED TREATMENT WITH NIVOLUMAB Patients who are found to have RECIST defined intracranial or extracranial progression (or both) from 6 weeks onwards, and who do not have clinical signs or symptoms of progression, may continue on nivolumab and must have a confirmatory scan within 4 to 6 weeks. The date of the original assessment of progression will be used to record progression, and not the date of the confirmatory imaging. Continued immunotherapy treatment is permitted if the treating clinician determines that the patient is still clinically benefiting from immunotherapy and the patient is willing to continue drug treatment. Consideration may be given to stable or good response extra- or intra- cranially with concurrent progression in the other as a scenario that may warrant further treatment.

There is growing evidence that patients may not need to be treated with immunotherapies indefinitely, or even for as long as the two years commonly studied in clinical trials. Rather, shorter courses of treatment may be just as effective and provide an option for retreatment should a patient progress after coming off a defined period of therapy. Patients who receive 2 years of immunotherapy have the option to cease treatment at this stage, with an option for a rechallenge of immunotherapy at the time of disease progression, if this occurs with 2 years of initial cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients, ≥18 years of age.
2. Signed, written, informed consent.
3. AJCC Stage IV [any T, any N, M1d (0) or M1D(1)] histologically confirmed cutaneous, acral or mucosal unresectable melanoma or unknown primary melanoma and at least 1 radiological definitive brain metastasis that is ≥ 5mm and ≤40mm, measurable per RECIST version 1.1 guidelines (modified for brain metastases, enabling up to 5 target lesions in the brain as well as up to 5 extracranial target lesions). There is no upper limit restriction in the number of brain metastases, provided the remaining eligibility criteria are met.
4. The BRAF mutation status must be available prior to randomisation.
5. The treating clinician(s) should consider the intracranial disease amenable to stereotactic radiotherapy over whole brain radiotherapy. Patients for whom there is a definite and immediate indication for radiotherapy (e.g. rapidly progressing disease with associated clinical signs and /or symptoms) should not be considered for enrolment.
6. Brain metastases must be untreated with any modality of radiotherapy or systemic treatment. Previous surgery for melanoma brain metastases is permitted if it resulted in gross total resection and no radiotherapeutic cavity boost was required.
7. No prior systemic treatment for brain metastases is permitted unless given in the neoadjuvant or adjuvant settings for systemic drug the treatment for extracranial disease only. At the time of neoadjuvant or adjuvant systemic therapy for extracranial disease, there should be radiological evidence of the absence of brain metastases. The presenting diagnosis of brain metastases at the time of enrolment in this study must have occurred a minimum of 6 months after stopping neoadjuvant or adjuvant systemic therapy (prior anti PD1, anti PD-L1, anti CTLA-4, BRAF / MEK inhibitors or clinical trial agents) are acceptable in the setting of neoadjuvant or adjuvant treatment
8. Asymptomatic from brain metastases at the time of study enrolment without corticosteroids, analgesia or any other treatment for the management of neurological symptoms (with the exception of antiepileptics prescribed for any reason, provided patient is asymptomatic). Resolved neurological symptoms are permitted if complete resolution, without any intervention, has been sustained for a minimum of 7 days prior to randomisation.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
10. A life expectancy > 30 days.
11. Able to undergo MRI with Gadolinium contrast agent. CT of the brain is not an acceptable alternative should patients be unable to safely undergo a contrast MRI.
12. Adequate haematological, hepatic and renal organ function as defined by:

    1. White cell count ≥ 2.0 × 10x9/L
    2. Neutrophil count ≥ 1.5 × 10x9/L
    3. Haemoglobin ≥ 90 g/L
    4. Platelet count ≥ 100 x 10x9/L
    5. Total bilirubin ≤ 1.5 x ULN
    6. Alanine transaminase ≤ 3.0 x ULN
    7. Aspartate aminotransferase ≤ 3.0 x ULN
    8. Serum creatinine ≤ 1.5 x the upper limit of normal (ULN). If serum creatinine is > 1.5 x ULN, calculate creatinine clearance using standard Cockcroft-Gault formula. Creatinine clearance must be 40ml/min to be eligible.
13. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first dose of study treatment and agree to use effective contraception from 14 days prior to commencing study treatment, throughout the treatment period and for 23 weeks * after the last dose of study treatment. Effective contraception includes:

    1. Intrauterine device with a documented failure rate of less than 1% per year.
    2. Vasectomised partner who is sterile prior to the female partner patient's commencement of study treatment and is the sole sexual partner for that female.
    3. Combined (oestrogen and progestogen) hormonal contraception associated with inhibition of ovulation or progestogen only hormonal contraception associated with inhibition of ovulation.

Women who are not of childbearing potential are defined as any female who has had a documented hysterectomy, bilateral oophorectomy or bilateral tubal ligation or any female who is post-menopausal (≥ one year without menses and >50 years of age in the absence of hormone replacement therapy).

* These durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days.

Exclusion Criteria

1. Patients whose intracranial disease changes between the diagnostic MRI scan and the baseline / SRS planning MRI scan and who are no longer suitable for SRS and / or require a specific alternative treatment outside of this protocol.
2. Melanoma brain metastasis greater than 40mm.
3. Evidence of leptomeningeal disease, with the exception of pathological findings seen at a previous resection of brain disease, but with no evidence of leptomeningeal disease elsewhere at the time of resection or at study entry.
4. History of, or current ocular melanoma (patients with mucosal and acral melanoma are eligible).
5. Neurological symptoms from brain metastases present at baseline (resolved neurological symptoms, prior to enrolment, are permitted).
6. Prior radiotherapy to the brain (surgery permitted).
7. Prior systemic drug therapy for melanoma, unless given in the neoadjuvant or adjuvant setting and completed 6 months before enrolment in this study.
8. Patients with active, known or suspected autoimmune disease. Patients with the following are permitted to enrol:

   1. Vitiligo
   2. Type I diabetes mellitus
   3. Residual hypothyroidism due to an autoimmune condition only requiring hormone replacement
   4. Psoriasis not requiring systemic treatment
   5. Autoimmune conditions not expected to recur in the absence of an external trigger.
9. Current systemic treatment with corticosteroids, or within 7 days of randomisation, with the exception of prednisone at non-immunosuppressive doses of ≤ 10 mg/day (or equivalent, e.g. e.g. prednisone 10mg = dexamethasone 1.6mg = hydrocortisone 40mg). Patients with the following circumstances are permitted to enrol:

   1. Past treatment for non-neurological symptoms allowed, if this was ceased 7 days prior to randomisation
   2. Inhaled or intranasal corticosteroids (with minimal systemic absorption) may be continued if the patient is on a stable dose
   3. Non-absorbed intra-articular steroid injections.

   During the study, treatment with systemic corticosteroids is permitted during radiotherapy if the patient experiences radiation related symptoms but this should be tapered per standard clinical practice as soon as possible and before the next infusion of study drug is due. This also refers to steroids for drug related signs or symptoms.
10. Any active infection requiring treatment.
11. A history of interstitial lung disease.
12. Any concurrent malignancy requiring any treatment or a history of another malignancy, unless the patient has been disease-free for 3 years.
13. Serious or unstable pre-existing medical conditions or other conditions that could interfere with the patient's safety, consent, or compliance.
14. Pregnant or breastfeeding females.
15. Administration of any form of live vaccine within 30 days of starting the trial and during the trial. Administration of any other vaccine is cautionary within 30 days of starting the trial and for the duration of the treatment phase of the trial.
16. Hypersensitivy to study treatments.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Neurological specific cause of death | One year
  Proportion of patients dead at one year from randomisation and whose immediate cause of death is neurological.

SECONDARY OUTCOMES:
Intracranial response rate | Up to 10 years
  The best response in intracranial metastases as measured using brain modified (bm) RECIST, following at least ONE dose of nivolumab and ipilimumab and based on imaging from week 6 onwards and confirmed a minimum of 4 weeks later.
Extracranial response rate | Approximately 10 years
  The best response in extracranial disease for each patient measured using bm RECIST, following at least ONE dose of nivolumab and ipilimumab and based on imaging from week 12 onwards.
Overall response rate | Up to 10 years
  Proportion of patients with an overall complete or partial response as measured using bm RECIST following at least ONE dose of nivolumab and ipilimumab and based on imaging from week 12 onwards .
Overall progression free survival | 1, 2, 5 and 10 years
  Time from the start of study treatment to the date of any progression of disease as measured using bm RECIST and based on imaging from week 12 onwards.
Non-Neurological specific cause of death | Up to 10 years
  Proportion of patients dead at one year from randomisation and whose immediate cause of death was due to melanoma but from causes other than brain metastases.
Overall survival | 1, 2, 5 and 10 years.
  Time from commencing study treatment to the date of death from any cause. Patients still alive at the end of the study will be censored at the date of their last assessment.
Incidence of radionecrosis | 5 years
  Proportion of patients with a diagnosis of radionecrosis occuring within 5 years of the start of the first course of radiotherapy.
Requirement for salvage radiotherapy | 1 year
  Proportion of patients requiring salvage radiotherapy in each cohort
Requirement for salvage intracranial surgery | 1 year
  Proportion of patients requiring salvage craniotomy in each cohort
Change in neurocognitive function scores | Up to 10 years
  The mean change from baseline assessment of neurocognitive function to the time of clinical response, stable disease and progression of disease.
Description of impaired neurological function and neurological adverse events | Up to 10 years
  Description of the nature of impaired function and types of neurological adverse events.
Time to neurological deterioration | Up to 10 years
  The time from starting immunotherapy to the time of deterioration of MoCA, CTCAE and FACT-Br.
Duration of neurological deterioration | Up to 10 years
  The time to resolution (if any) of each functional neurocognitive deficit.
Patient rated quality of life | Up to 10 years
  Time from starting study treatment to the time of deterioration in quality life scores and the duration of deterioration.
Functional performance status | Up to 10 years
  Incidence of reduced functional performance by 1, 2 or 3 grades of the Eastern Cooperative Oncology Group (ECOG) performance status scale compared to baseline.
Adverse events | Up to 10 years
  Description of all adverse events per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Tissue, blood and gut biomarkers of response, progression and toxicity | Up to 10 years
  Correlation of the baseline PD-L1 status, immune markers, genomics and other biomarkers in tumour tissue and blood and the composition and diversity of the gut microbiome with RECIST response and toxicity. Correlation of gastrointestinal mucosal integrity with bacterial composition in stool samples, RECIST response and immune related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Georgina V Long, MBBS PhD, Study Chair — Melanoma Institute Australia
Locations (9):
- Australia (8):
  - Westmead Hospital, Sydney, New South Wales
  - Calvary Mater NewcastleHospital, Waratah, New South Wales
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hosptial, Perth, Western Australia
- Oslo Univesity Hospital Radiumhospitalet, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phillips WJ, Baghai T, Ong M, Lo B, Ibrahim AM, Smith TKT, Song X. A Contemporary Report of Clinical Outcomes in Patients with Melanoma Brain Metastases. Curr Oncol. 2021 Jan 13;28(1):428-439. doi: 10.3390/curroncol28010045. PMID 33450821
- See also: Trial Information — https://melanoma.org.au/research/clinical-trials/abc-x-clinical-trial/